CLINICAL TRIAL: NCT05921435
Title: A Phase I Clinical Trial to Compare and Evaluate the Safety and Pharmacokinetic Characteristics After Administration of D958 and CKD-341 in Healthy Adult Volunteers
Brief Title: Clinical Trial to Compare and Evaluate the Safety and Pharmacokinetic After Oral Administration of CKD-341 and D958 in Healthy Adults
Acronym: CKD-341
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A126_02BE2303
Record Dates: First submitted 2023-06-18; First posted 2023-06-27 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2023-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): * Period 1: D958
  * Period 2: CKD-341
  * Period 3: D958
  * Period 4: CKD-341
  Interventions: Drug: CKD-341, D958
- Sequence B (Experimental): * Period 1: CKD-341
  * Period 2: D958
  * Period 3: CKD-341
  * Period 4: D958
  Interventions: Drug: CKD-341, D958

INTERVENTIONS:
Drug: CKD-341, D958 — A single dose of 1tablet under fasting condition

SUMMARY:
A clinical trial to compare and evaluate the safety and pharmacokinetics of CKD-341

DETAILED DESCRIPTION:
A Randomized, Open-label, Oral, Single-dose, 2-treatment, Replicate crossover, 4-period Stuy

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult subjects aged over 19 years (inclusive) at the time of screening.
2. Subjects weighing at least 50.0 kg with a Body Mass Index(BMI) between 18.0 kg/m2 and 30.0 kg/m2 (inclusive) at the time of screening.

   * BMI(kg/m2) = weight (kg) / {height (m)}2
3. Subjects with neither congenital nor chronic diseases requiring treatment, and no abnormal symptoms or findings upon medical examination.
4. Subjects considered eligible for the study participation in accordance with the results of vital signs, physical examination, 12-lead ECG, and clinical laboratory tests at the time of screening.
5. Subjects who have a full understanding in participation of the study, voluntarily provide a written consent in participation, and give full agreement in following the subject guidelines throughout the entire study period.

Exclusion Criteria:

1. Subjects with any clinically significant past and present hepatic, renal, nervous, respiratory, endocrine, circulatory, oncologic, genitourinary, cardiovascular, digestive, musculoskeletal systemic diseases, psychosis disorders, or a medical history of at least one of the following conditions (past and present):

   1-1) Liver disorders and biliary obstructive disease 1-2) Kidney disorders 1-3) Shock 1-4) Hypokalemia, hyponatremia, hypercalcemia 1-5) Addison's syndrome 1-6) Primary aldosteronism 1-7) Aortic stenosis, mitral obstruction or hypertrophic obstructive cardiomyopathy 1-8) Renovascular hypertension or anuria 1-9) Hypotension 1-10) Vascular sclerosis or cerebral arteriosclerosis 1-11) Hyperuricemia (with gout or uric acid stone) or diabetes (including family history) 1-12) Hyperparathyroidism 1-13) Sympathectomy
2. For women, pregnant (urine-HCG positive) or lactating women
3. History of any clinically significant hypersensitivity reactions or hypersensitivity reactions to any of the IP main ingredients, formulation additives, and other drugs (including dihydropyridine derivatives, thiazide diuretics, or sulfonamide drugs).
4. Subjects on lithium therapy or salt-restricted therapy
5. Subjects with hereditary issues of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption, etc.
6. Subjects with a past medical history of gastrointestinal disease (Crohn's disease, ulcers, acute/chronic pancreatitis, etc.) or gastrointestinal surgeries (except for simple appendectomy and hernia repair) which may affect the absorption of the IP.
7. Subjects with clinically significant 12-lead ECG findings including the following results at the time of screening:

   * QTc > 450 ms for men, QTc > 470 ms for women
   * PR interval > 200 ms
   * QRS duration > 120 ms
8. Subjects with laboratory test results as follows at the time of screening:

   * Liver function test (AST, ALT, ALP, γ-GTP and total bilirubin) values exceeding twice the upper normal limit
   * Creatinine values outside the reference ranges or eGFR < 60 mL/min/1.73m2 (eGFR is estimated using the Chronic Kidney Disease Epidemiology Collaboration formula)
   * CPK > 2.5 times the upper limit of normal range on clinical laboratory tests
9. Subjects with a past history of drug abuse or a positive urine drug screening test
10. Subjects with systolic blood pressure ≥ 150 mmHg or ≤ 90 mmHg; diastolic blood pressure ≥ 100 mmHg or ≤ 60 mmHg; pulse rate ≤ 40 beats/min or ≥ 100 beats/min, when measured in a seated position without an abrupt change in body position for at least 3 minutes at the time of screening
11. Subjects taking drugs known to significantly induce or inhibit drug metabolizing enzymes, including barbitals, within 1 month prior to the first IP administration
12. Subjects following an unusual diet or consumption of food which may affect the absorption, distribution, metabolism and excretion of the IP
13. Subjects who have taken any prescribed medications including cyclosporine, nonsteroidal anti-inflammatory drugs, terfenadine, astemizole, digitalis, glucocorticoids, adrenocorticotropic hormone, and agents that affect the renin-angiotensin-aldosterone system (RAAS) or herbal medicine within 2 weeks or any over-the-counter drug or vitamin supplements within 10 days prior to the first IP administration (except for circumstances considered acceptable with no concerned effect on the pharmacokinetics (PK) of the IP at the investigator's discretion)
14. Subjects who have participated and were given any other study drugs in other clinical study within 6 months prior to the first IP administration (the last day of IP administration is considered the end-of-study)
15. Subjects who have donated whole blood within 2 months or blood components within 1 month or received a blood transfusion within 1 month prior to the first IP administration or subjects unable to abstain from donating blood from the time of consent until PSV
16. Subjects who have consistently drunk alcohol within 6 months exceeding 21 units/week (1 unit = 10 g = 12.5 mL of pure alcohol) prior to the first IP administration or are unable to refrain from drinking from the time of consent until PSV
17. Subjects who have smoked more than 10 cigarettes/day on average 3 months prior to the first IP administration and are unable to oblige the no-smoking rules from 24 hours prior to IP administration until the last blood sampling point for each period
18. Subjects who have consumed and are unable to refrain from consuming grapefruit-containing food or beverages from 48 hours prior to the first IP administration until PSV
19. Subjects who have consumed and are unable to refrain from consuming caffeine-containing food or beverages (coffee, green tea, black tea, carbonated drinks, coffee-flavored milk, energy drinks, etc.) from 24 hours prior to IP administration until the last blood sampling point for each period
20. Subjects who have done and are unable to refrain from strenuous activity from 48 hours prior to the first IP administration until PSV
21. Subjects who are planning for pregnancy or not willing to use a medically reliable forms of contraception (administration of contraceptives or transplantation of contraceptives or use of an intrauterine device, steriliaztion surgery (vasectomy or tubal ligation), and physical barriers (spermicide, condom, contraceptive diaphragm, vaginal sponge used with a cervical cap)) from the time of consent until 2 weeks after the last IP administration
22. Subjects otherwise considered ineligible for participation due to other reasons not mentioned in the inclusion/exclusion criteria at the investigator's discretion

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 48 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
area under curve(AUC) of CKD-341, D958 | Pre-dose(0 hour), post-dose 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72, 96, 144 hours
  Area under the CKD-341, D958 concentration in blood-time curve from zero to final
Cmax of CKD-341, D958 | Pre-dose(0 hour), post-dose 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72, 96, 144 hours
  The maximum CKD-341, D958 concentration in blood sampling time

CONTACTS AND LOCATIONS:
Locations (1):
- Chungbuk National University Hospital, Cheongju-si, South Korea

IPD SHARING:
Plan to Share IPD: No